CLINICAL TRIAL: NCT03265938
Title: Evaluation of Video Laryngoscopy in Patients With Head and Neck Pathology
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jaime B Hyman, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 17-0963
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Difficult Intubation
Keywords: Head and Neck cancer; Cancer of oral cavity; Ear, Nose and Throat; Indirect laryngoscopy; Awake intubation; Expected difficult intubation
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Indirect laryngoscopy: Head and neck pathology patients undergoing indirect laryngoscopy. Patients with a past medical history of active or previously treated head and neck pathology.
  Interventions: Device: Indirect Laryngoscopy

INTERVENTIONS:
Device: Indirect Laryngoscopy — The attending anesthesiologist will perform video laryngoscopy with the C-MAC D video laryngoscope and with the GlideScope AVL video laryngoscope and grade the view of the larynx obtained with each laryngoscope.
  Other Names: Glidescope AVL Indirect Laryngoscopy; C-MAC D-Blade Indirect Laryngoscopy

SUMMARY:
Patients who undergo general anesthesia for surgical procedures frequently need to have a breathing tube placed ("tracheal intubation") for the duration of the procedure. Most often airway management is routine for an experienced anesthesiologist. Less often, airway management can be difficult and can result in patient harm. In order to reduce risk, anesthesiologists routinely evaluate patients' airways by obtaining a relevant history and doing a physical exam, which can aid in predicting which airways may be difficult to manage. The "gold standard" for management of the anticipated difficult airway is to perform an awake flexible bronchoscopic intubation after anesthetizing the airway with local anesthesia. This affords added safety because the airway remains patent and the patient breaths spontaneously until a tracheal tube is secured, at which point general anesthesia can be induced.

Recently, authors have advocated for alternative methods of management of the predicted difficult airway, most commonly by using a video laryngoscope to perform the awake intubation. A video laryngoscope provides an indirect view of the larynx using a camera at the tip of a rigid laryngoscope. It takes less training to gain and maintain proficiency compared to flexible bronchoscopy.

Previous studies that have shown successful awake intubation with video laryngoscopy in the predicted difficult airway have not included patients with head and neck pathology, including malignancies or a history of head and neck surgery or radiation. In this study, the study team will perform video laryngoscopy in patients with head and neck pathology who require awake bronchoscopic intubation for surgery after placement of the tracheal tube and induction of anesthesia. The study team hypothesize that it will be difficult to obtain a good view of the larynx with video laryngoscopy in some patients with head and neck pathology. If there is a significant incidence of difficult video laryngoscopy in this patient population, it will reinforce that anesthesiologists need to continue to learn and maintain skills in bronchoscopic intubation.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* Presence of oral, pharyngeal or laryngeal mass or history of surgery or radiation for head and neck cancer
* Requiring awake flexible bronchoscopic intubation for surgery
* Willing and able to provide informed consent

Exclusion Criteria:

* Emergency Procedure
* Presence of one or more loose teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all patients scheduled to undergo a surgical procedure at the Mount Sinai Hospital (New York, NY)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Hyman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apfelbaum JL, Hagberg CA, Caplan RA, Blitt CD, Connis RT, Nickinovich DG, Hagberg CA, Caplan RA, Benumof JL, Berry FA, Blitt CD, Bode RH, Cheney FW, Connis RT, Guidry OF, Nickinovich DG, Ovassapian A; American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2013 Feb;118(2):251-70. doi: 10.1097/ALN.0b013e31827773b2. No abstract available. PMID 23364566
- [Background] Ahmad I, Bailey CR. Time to abandon awake fibreoptic intubation? Anaesthesia. 2016 Jan;71(1):12-6. doi: 10.1111/anae.13333. No abstract available. PMID 26684527
- [Background] Kramer A, Muller D, Pfortner R, Mohr C, Groeben H. Fibreoptic vs videolaryngoscopic (C-MAC((R)) D-BLADE) nasal awake intubation under local anaesthesia. Anaesthesia. 2015 Apr;70(4):400-6. doi: 10.1111/anae.13016. PMID 25764403
- [Background] Rosenstock CV, Thogersen B, Afshari A, Christensen AL, Eriksen C, Gatke MR. Awake fiberoptic or awake video laryngoscopic tracheal intubation in patients with anticipated difficult airway management: a randomized clinical trial. Anesthesiology. 2012 Jun;116(6):1210-6. doi: 10.1097/ALN.0b013e318254d085. PMID 22487805
- [Background] Aziz MF, Healy D, Kheterpal S, Fu RF, Dillman D, Brambrink AM. Routine clinical practice effectiveness of the Glidescope in difficult airway management: an analysis of 2,004 Glidescope intubations, complications, and failures from two institutions. Anesthesiology. 2011 Jan;114(1):34-41. doi: 10.1097/ALN.0b013e3182023eb7. PMID 21150569
- [Background] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Background] Fiadjoe JE, Litman RS. Difficult tracheal intubation: looking to the past to determine the future. Anesthesiology. 2012 Jun;116(6):1181-2. doi: 10.1097/ALN.0b013e318254d0a0. No abstract available. PMID 22487804
- [Background] Popat MT, Srivastava M, Russell R. Awake fibreoptic intubation skills in obstetric patients: a survey of anaesthetists in the Oxford region. Int J Obstet Anesth. 2000 Apr;9(2):78-82. doi: 10.1054/ijoa.1999.0361. PMID 15321093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: study was conducted from September 2017 until July 2019
Groups:
- Indirect Laryngoscopy: Head and neck pathology patients undergoing indirect laryngoscopy. Indirect Laryngoscopy: The attending anesthesiologist will perform video laryngoscopy with the C-MAC D video laryngoscope and with the GlideScope AVL video laryngoscope and grade the view of the larynx obtained with each laryngoscope.
Period: Overall Study
Arm/Group | Indirect Laryngoscopy
Started | 100
Completed | 92
Not Completed | 8
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — friable mass | 6

BASELINE CHARACTERISTICS:
Arm/Group | Indirect Laryngoscopy
Number analyzed (Participants) | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [56.25 to 71.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 75
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 23.79 [21.67 to 27.46]
History of Head and Neck Surgery [Count of Participants; unit: Participants] | 49
History of Radiation Therapy [Count of Participants; unit: Participants] | 69
Edentulous [Count of Participants; unit: Participants] | 25
Mallampati score [Count of Participants; unit: Participants] — the Mallampati score (or Mallampati classification) is used to predict the ease of intubation.
  1. Complete visualization of the soft palate
  2. Complete visualization of the uvula
  3. Visualization of only the base of the uvula
  4. Soft palate is not visible at all
  Participants
    1 | 8
    2 | 32
    3 | 24
    4 | 36
Head and Neck Mass Location [Count of Participants; unit: Participants]
  None | 45
  Base of Tongue | 23
  Supraglottic | 11
  Neck | 11
  Laryngeal | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cormack-Lehane Grade >2 Obtained With CMAC D Blade
Description: Number of participants with difficult (Cormack-Lehane grade >2) video laryngoscopic view of the larynx after awake flexible bronchoscopic intubation in patients with head and neck pathology with CMAC
  Cormack-Lehane grade in patients with head and neck pathology of the larynx.
  Cormack-Lehane grade:
  Grade 1: full view of the glottis Grade 2a: partial view of the glottis Grade 2b: arytenoids only Grade 3: epiglottis only Grade 4: neither glottis or epiglottis identified
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- Indirect Laryngoscopy: Head and neck pathology patients undergoing indirect laryngoscopy. Indirect Laryngoscopy: The attending anesthesiologist performed video laryngoscopy with the C-MAC D video laryngoscope and graded the view of the larynx.
Arm/Group | Indirect Laryngoscopy
Number analyzed (Participants) | 92
Participants | 37

2. Primary Outcome: Number of Participants With Cormack-Lehane Grade >2 Obtained With Glidescope AVL
Description: Number of participants with difficult (Cormack-Lehane grade >2) video laryngoscopic view of the larynx after awake flexible bronchoscopic intubation in patients with head and neck pathology obtained with Glidescope AVL
  Cormack-Lehane grade in patients with head and neck pathology of the larynx.
  Cormack-Lehane grade:
  Grade 1: full view of the glottis Grade 2a: partial view of the glottis Grade 2b: arytenoids only Grade 3: epiglottis only Grade 4: neither glottis or epiglottis identified
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- Indirect Laryngoscopy: Head and neck pathology patients undergoing indirect laryngoscopy. Indirect Laryngoscopy: The attending anesthesiologist performed video laryngoscopy with the GlideScope AVL video laryngoscope and graded the view of the larynx.
Arm/Group | Indirect Laryngoscopy
Number analyzed (Participants) | 92
Participants | 28

3. Secondary Outcome: Cormack-Lehane Grade Obtained With CMAC D Blade
Description: Cormack-Lehane grade in patients with head and neck pathology of the larynx.
  Cormack-Lehane grade:
  Grade 1: full view of the glottis Grade 2a: partial view of the glottis Grade 2b: arytenoids only Grade 3: epiglottis only Grade 4: neither glottis or epiglottis identified
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Indirect Laryngoscopy
Number analyzed (Participants) | 92
Participants
  Grade 1 | 23
  Grade 2a | 19
  Grade 2b | 13
  Grade 3 | 8
  Grade 4 | 29

4. Secondary Outcome: Cormack-Lehane Grade Obtained With Glidescope AVL
Description: as for outcome 3
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Indirect Laryngoscopy
Number analyzed (Participants) | 92
Participants
  Grade 1 | 37
  Grade 2a | 14
  Grade 2b | 13
  Grade 3 | 6
  Grade 4 | 22

5. Secondary Outcome: Cormack-Lehane Grade in Patients With Head and Neck Masses Obtained With CMAC D Blade
Description: Cormack-Lehane view obtained by video laryngoscopy after awake flexible bronchoscopic intubation in patients with head and neck masses.
Time Frame: Day 1
Population: Data for participants who have a history of head and neck masses.
Measure: Count of Participants; unit: Participants
Arm/Group | Indirect Laryngoscopy
Number analyzed (Participants) | 48
Participants
  Grade 1 | 11
  Grade 2a | 10
  Grade 2b | 8
  Grade 3 | 4
  Grade 4 | 15

6. Secondary Outcome: Cormack-Lehane Grade in Patients With Head and Neck Masses Obtained With Glidescope AVL
Description: as for outcome 5
Time Frame: Day 1
Population: Data for participants who have a history of head and neck masses.
Measure: Count of Participants; unit: Participants
Arm/Group | Indirect Laryngoscopy
Number analyzed (Participants) | 48
Participants
  Grade 1 | 19
  Grade 2a | 5
  Grade 2b | 10
  Grade 3 | 2
  Grade 4 | 12

7. Secondary Outcome: Cormack-Lehane Grade in Patients With Neck Radiation Obtained With CMAC D Blade
Description: Cormack-Lehane view obtained by video laryngoscopy after awake flexible bronchoscopic intubation in patients with a history of neck radiation.
Time Frame: Day 1
Population: Data for participants who have a history of neck radiation
Measure: Count of Participants; unit: Participants
Arm/Group | Indirect Laryngoscopy
Number analyzed (Participants) | 66
Participants
  Grade 1 | 18
  Grade 2a | 10
  Grade 2b | 9
  Grade 3 | 6
  Grade 4 | 23

8. Secondary Outcome: Cormack-Lehane Grade in Patients With Neck Radiation Obtained With Glidescope AVL
Description: as for outcome 7
Time Frame: Day 1
Population: Data for participants who have a history of neck radiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Indirect Laryngoscopy
Number analyzed (Participants) | 66
Participants
  Grade 1 | 26
  Grade 2a | 11
  Grade 2b | 9
  Grade 3 | 5
  Grade 4 | 15

ADVERSE EVENTS:
Time Frame: 1 Day
Arm/Group | Indirect Laryngoscopy
All-Cause Mortality (participants affected / at risk) | 0/92
Serious Adverse Events (participants affected / at risk) | 0/92
Other Adverse Events (participants affected / at risk) | 0/92

LIMITATIONS AND CAVEATS:
This study was not a comparison between awake techniques. Laryngoscopy conditions may be different after an endotracheal tube is already in place and the patient is anesthetized. The results cannot be generalized to other available types.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT03265938/Prot_SAP_000.pdf